CLINICAL TRIAL: NCT00045162
Title: Randomized Phase III Trial of Cisplatin and Irinotecan (NSC-616348) Versus Cisplatin and Etoposide in Patients With Extensive Stage Small Cell Lung Cancer (E-SCLC)
Brief Title: S0124: Cisplatin Combined With Irinotecan or Etoposide For Extensive-Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH); North Central Cancer Treatment Group (Network); Cancer and Leukemia Group B (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000256908; S0124 (Other: SWOG); S0124 (Other: NCCTG); S0124 (Other: CALGB); U10CA032102 (NIH)
Record Dates: First submitted 2002-09-06; First posted 2003-01-27 (Estimated); Results first posted 2013-07-09 (Estimated); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Lung Cancer
Keywords: extensive stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Cisplatin; Etoposide; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: cisplatin; Drug: irinotecan hydrochloride
- 2 (Active Comparator)
  Interventions: Drug: cisplatin; Drug: etoposide

INTERVENTIONS:
Drug: cisplatin — Arm 1: 60 mg/m2 IV (over 30-60 min) on Day 1, Q 4 weeks x 4 Cycles
  Arm 2: 80 mg/m2 IV (over 30-60 min) on Day 1, Q 4 weeks x 4 Cycles
Drug: etoposide — 100 mg/m2 IV (over 30-60 min) on Days 1 , 2 & 3. Q 3 weeks x 4 Cycles
  Arms: 2
Drug: irinotecan hydrochloride — 60 mg/m2 IV (over 90 min)on Days 1, 8 & 15. Q 4 weeks x 4 Cycles
  Arms: 1

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known whether cisplatin combined with irinotecan is more effective than cisplatin combined with etoposide in treating extensive-stage small cell lung cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of cisplatin combined with either irinotecan or etoposide in treating patients who have extensive-stage small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the survival of patients with extensive stage small cell lung cancer treated with cisplatin and irinotecan vs cisplatin and etoposide.
* Compare the objective response rate and progression-free survival of patients treated with these regimens.
* Compare the toxic effects of these regimens in these patients.
* Determine the association between UGT1A1 polymorphisms and irinotecan-associated toxic effects in these patients.
* Determine the association between ERCC-1 and XRCC-1 polymorphisms and non-response of patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to number of metastatic sites (single vs multiple), lactic dehydrogenase (no greater than upper limit of normal (ULN) vs greater than ULN), and weight loss in the past 6 months (5% or less vs more than 5%). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive irinotecan IV over 90 minutes on days 1, 8, and 15 and cisplatin IV over 30-60 minutes on day 1. Courses repeat every 4 weeks.
* Arm II: Patients receive etoposide IV over 30-60 minutes on days 1-3 and cisplatin IV over 30-60 minutes on day 1. Courses repeat every 3 weeks.

Treatment in both arms continues for 4 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 1 year and then every 6 months for 2 years.

PROJECTED ACCRUAL: A total of 620 patients (310 per treatment arm) will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed extensive stage small cell lung cancer (SCLC)
* Measurable or evaluable disease by CT scan, MRI, x-ray, physical exam, or nuclear exam
* Brain metastases allowed if previously treated with radiotherapy and/or surgery and are neurologically stable (i.e., no progressing symptoms and off steroids and anticonvulsants)

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Zubrod 0-1

Life expectancy

* Not specified

Hematopoietic

* WBC at least 3,000/mm^3
* Absolute granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST or ALT no greater than 2.5 times ULN

Renal

* Creatinine normal
* Creatinine clearance at least 50 mL/min

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* HIV negative
* No concurrent AIDS-related illness

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior biologic therapy for SCLC
* No filgrastim (G-CSF) within 24 hours of chemotherapy

Chemotherapy

* No prior systemic chemotherapy for SCLC

Endocrine therapy

* See Disease Characteristics

Radiotherapy

* See Disease Characteristics
* At least 21 days since prior brain radiotherapy and recovered
* No other prior radiotherapy for SCLC

Surgery

* See Disease Characteristics
* At least 21 days since prior thoracic or other major surgery and recovered

Other

* No concurrent enzyme inducing antiepileptic drugs (phenytoin, phenobarbital, oxcarboxepine, or carbamazepine)

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 671 (Actual)
Dates: Start 2002-11; Primary Completion 2008-03 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald B. Natale, MD, Principal Investigator — Cedars-Sinai Medical Center; David R. Gandara, MD, Principal Investigator — University of California, Davis; Primo N. Lara, MD, Principal Investigator — University of California, Davis; James R. Jett, MD, Principal Investigator — Mayo Clinic; Jane Carleton, MD, Principal Investigator — Don Monti Comprehensive Cancer Center at North Shore University Hospital
Locations (408):
- United States (406):
  - Northeast Alabama Regional Medical Center, Anniston, Alabama
  - Huntsville Hospital, Huntsville, Alabama
  - Mobile Infirmary Medical Center, Mobile, Alabama
  - East Alabama Medical Center, Opelika, Alabama
  - Alaska Regional Hospital Cancer Center, Anchorage, Alaska
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Hembree Mercy Cancer Center at St. Edward Mercy Medical Center, Fort Smith, Arkansas
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Providence Saint Joseph Medical Center - Burbank, Burbank, California
  - Cancer Care Center at John Muir Health - Concord Campus, Concord, California
  - Washington Township Hospital, Fremont, California
  - California Cancer Center - Woodward Park Office, Fresno, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Desert Regional Medical Center Comprehensive Cancer Center, Palm Springs, California
  - Shasta Regional Medical Center, Redding, California
  - Sutter Cancer Center at Roseville Medical Center, Roseville, California
  - Sutter Cancer Center, Sacramento, California
  - University of California Davis Cancer Center, Sacramento, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - John Muir/Mt. Diablo Comprehensive Cancer Center, Walnut Creek, California
  - Memorial Hospital, Colorado Springs, Colorado
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Halifax Medical Center - Daytona Beach, Daytona Beach, Florida
  - Broward General Medical Center Cancer Center, Fort Lauderdale, Florida
  - West Florida Cancer Institute at West Florida Hospital - Pensacola, Pensacola, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Northside Hospital Cancer Center, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Augusta Oncology Associates - Walton Way, Augusta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - Charles B. Eberhart Cancer Center at DeKalb Medical Center, Decatur, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Kennestone Cancer Center at Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Curtis & Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Pearlman Comprehensive Cancer Center at South Georgia Medical Center, Valdosta, Georgia
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Hematology Oncology Associates of Eastern Idaho, Idaho Falls, Idaho
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Veterans Affairs Medical Center - Hines, Hines, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - La Grange Memorial Hospital, La Grange, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Trinity Medical Center - East, Moline, Illinois
  - Moline, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - West Suburban Center for Cancer Care, River Forest, Illinois
  - Swedish-American Regional Cancer Center, Rockford, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital at Howard Regional Health System, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Reid Hospital & Health Care Services, Incorporated, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Bettendorf, Iowa
  - St. Luke's Hospital, Cedar Rapids, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Heartland Oncology & Hematology, Council Bluffs, Iowa
  - Genesis Regional Cancer Center at Genesis Medical Center, Davenport, Iowa
  - Genesis Medical Center - West Campus, Davenport, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cedar Valley Medical Specialists, PC - West Ridgeway Avenue, Waterloo, Iowa
  - Covenant Cancer Treatment Center, Waterloo, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Tammy Walker Cancer Center at Salina Regional Health Center, Salina, Kansas
  - Stormont-Vail Cancer Center, Topeka, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Merle M. Mahr Cancer Center at Regional Medical Center of Hopkins County, Madisonville, Kentucky
  - Tulane Cancer Center, Alexandria, Louisiana
  - Louisiana State University Health Sciences Center - Monroe, Monroe, Louisiana
  - Christus Schumpert Cancer Treatment Center, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Feist-Weiller Cancer Center at Louisiana State University Health Sciences, Shreveport, Louisiana
  - CancerCare of Maine at Eastern Maine Medial Center, Bangor, Maine
  - MaineGeneral Medical Center - Waterville Campus, Waterville, Maine
  - Sturdy Memorial Hospital, Attleboro, Massachusetts
  - Cancer Research Center at Boston Medical Center, Boston, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - UMASS Memorial Cancer Center - University Campus, Worcester, Massachusetts
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Spectrum Health Hospital - Butterworth Campus, Grand Rapids, Michigan
  - Metro Health Hospital, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Green Bay Oncology, Limited - Iron Mountain, Iron Mountain, Michigan
  - Foote Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - Upper Michigan Cancer Center at Marquette General Hospital, Marquette, Michigan
  - MidMichigan Medical Center - Midland, Midland, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital System, Monroe, Michigan
  - Ted B. Wahby Cancer Center at Mount Clemens General Hospital, Mount Clemens, Michigan
  - Hackley Hospital, Muskegon, Michigan
  - Northern Michigan Hospital, Petoskey, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute - Saginaw, Saginaw, Michigan
  - Lakeland Cancer Care Center at Lakeland Hospital - St. Joseph, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Alexandria, Minnesota
  - MeritCare Clinic - Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Cancer Care Center at St. Luke's Hospital, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller-Dwan Medical Center, Duluth, Minnesota
  - St. Mary's - Duluth Clinic Cancer Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Fergus Falls, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - Immanuel St. Joseph's Clinic, Mankato, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA at Maplewood Cancer Center, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Chippewa County - Montevideo Hospital, Montevideo, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Medical Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Health Services, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - St. Joseph's Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Cancer Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Woodwinds Health Campus, Woodbury, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Missouri Regional Cancer Center at Southeast Missouri Hospital, Cape Girardeau, Missouri
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Capital Region Cancer Center, Jefferson City, Missouri
  - Freeman Cancer Institute at Freeman Health System, Joplin, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Arch Medical Services, Incorporated at Center for Cancer Care Research, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare, Billings, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Deaconess Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Community Hospital, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Sletten Regional Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Methodist Cancer Center at Methodist Hospital - Omaha, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Hunterdon Regional Cancer Center at Hunterdon Medical Center, Flemington, New Jersey
  - Carol G. Simon Cancer Center at Morristown Memorial Hospital, Morristown, New Jersey
  - Jersey Shore Cancer Center at Jersey Shore University Medical Center, Neptune City, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Finger Lakes Hematology and Oncology, Clifton Springs, New York
  - Adirondack Cancer Care - Glens Falls, Glens Falls, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Don Monti Comprehensive Cancer Center at North Shore University Hospital, Manhasset, New York
  - Tucker Center for Cancer Care at Orange Regional Medical Center, Middletown, New York
  - Winthrop University Hospital, Mineola, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Interlakes Oncology/Hematology PC, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Lenoir Memorial Cancer Center, Kinston, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Zimmer Cancer Center at New Hanover Regional Medical Center, Wilmington, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - Dakota Cancer Institute at Dakota Clinic - South University, Fargo, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Wood County Oncology Center, Bowling Green, Ohio
  - Mercy Cancer Center at Mercy Medical Center, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - MetroHealth's Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Riverside Cancer Services, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Fremont Memorial Hospital, Fremont, Ohio
  - Community Oncology Group at Cleveland Clinic Cancer Center, Independence, Ohio
  - Kenton Oncology, Incorporated, Kenton, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - MedCentral - Mansfield Hospital, Mansfield, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - Middletown Regional Hospital, Middletown, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Mount Carmel Cancer Services at Mount Carmel St. Ann's Hospital, Westerville, Ohio
  - Cleveland Clinic - Wooster, Wooster, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Tod Children's Hospital - Forum Health, Youngstown, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Merle West Medical Center Cancer Treatment Center, Klamath Falls, Oregon
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - Kaiser Permanente Health Care - Portland, Portland, Oregon
  - Oregon Health & Science University Cancer Institute, Portland, Oregon
  - Salem Hospital Regional Cancer Care Services, Salem, Oregon
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Oncology Hematology Associates of Northern Pennsylvania, PC at Hahne Regional Cancer Center, DuBois, Pennsylvania
  - Easton Regional Cancer Center at Easton Hospital, Easton, Pennsylvania
  - PinnacleHealth Regional Cancer Center at Polyclinic Hospital, Harrisburg, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - St. Mary Regional Cancer Center, Langhorne, Pennsylvania
  - Allegheny Cancer Center at Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - Hematology and Oncology Associates of Northeastern Pennsylvania, Scranton, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - AnMed Cancer Center, Anderson, South Carolina
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Bon Secours St. Francis Health System, Greenville, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - U.T. Cancer Institute at University of Tennessee Medical Center, Knoxville, Tennessee
  - University of Tennessee Cancer Institute - Medical Center, Memphis, Tennessee
  - Medical City Dallas Hospital, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Baylor University Medical Center - Houston, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Methodist Hospital, Houston, Texas
  - St. Luke's Texas Cancer Institute at St. Luke's Episcopal Hospital, Houston, Texas
  - Veterans Affairs Medical Center - Houston, Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - UMC Southwest Cancer and Research Center, Lubbock, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Cancer Therapy and Research Center, San Antonio, Texas
  - University Hospital - San Antonio, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - American Fork Hospital, American Fork, Utah
  - Logan Regional Hospital, Logan, Utah
  - Cottonwood Hospital Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - Latter Day Saints Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Martha Jefferson Hospital Cancer Care Center, Charlottesville, Virginia
  - Danville Regional Medical Center, Danville, Virginia
  - Lynchburg Hematology-Oncology Clinic, Lynchburg, Virginia
  - Peninsula Cancer Institute - Newport News Office, Newport News, Virginia
  - Veterans Affairs Medical Center - Richmond, Richmond, Virginia
  - Auburn Regional Center for Cancer Care, Auburn, Washington
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Providence Centralia Hospital Regional Cancer Center, Centralia, Washington
  - St. Francis Hospital, Federal Way, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Providence St. Peter Hospital Regional Cancer Center, Olympia, Washington
  - Good Samaritan Cancer Center, Puyallup, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Rockwood Clinic Cancer Treatment Center, Spokane, Washington
  - Providence Cancer Center at Sacred Heart Medical Center, Spokane, Washington
  - Providence Cancer Center at Holy Family Hospital, Spokane, Washington
  - St. Joseph Medical Center at Franciscan Health System, Tacoma, Washington
  - Allenmore Hospital, Tacoma, Washington
  - CCOP - Northwest, Tacoma, Washington
  - MultiCare Regional Cancer Center at Tacoma General Hospital, Tacoma, Washington
  - St. Clare Hospital, Tacoma, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Fox Valley Hematology and Oncology - East Grant Street, Appleton, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Mercy Regional Cancer Center, Janesville, Wisconsin
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - All Saints Cancer Center at Wheaton Franciscan Healthcare, Racine, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - University of Wisconcin Cancer Center at Aspirus Wausau Hospital, Wausau, Wisconsin
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming
- Canada (2):
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan
  - Saskatoon Cancer Centre at the University of Saskatchewan, Saskatoon, Saskatchewan

REFERENCES:
- [Background] Lara P, Chansky K, Shibata T, et al.: Cisplatin + irinotecan versus cisplatin + etoposide in extensive stage small cell lung cancer (E-SCLC): Final "common arm": comparative outcomes analysis of JCOG 9511 and SWOG 0124. [Abstract] J Clin Oncol 27 (Suppl 15): A-8027, 2009.
- [Result] Lara PN Jr, Natale R, Crowley J, Lenz HJ, Redman MW, Carleton JE, Jett J, Langer CJ, Kuebler JP, Dakhil SR, Chansky K, Gandara DR. Phase III trial of irinotecan/cisplatin compared with etoposide/cisplatin in extensive-stage small-cell lung cancer: clinical and pharmacogenomic results from SWOG S0124. J Clin Oncol. 2009 May 20;27(15):2530-5. doi: 10.1200/JCO.2008.20.1061. Epub 2009 Apr 6. PMID 19349543
- [Result] Natale RB, Lara PN, Chansky K, et al.: S0124: A randomized phase III trial comparing irinotecan/cisplatin (IP) with etoposide/cisplatin (EP) in patients (pts) with previously untreated extensive stage small cell lung cancer (E-SCLC). [Abstract] J Clin Oncol 26 (Suppl 15): A-7512, 2008.
- [Result] Hanna N, Bunn PA Jr, Langer C, Einhorn L, Guthrie T Jr, Beck T, Ansari R, Ellis P, Byrne M, Morrison M, Hariharan S, Wang B, Sandler A. Randomized phase III trial comparing irinotecan/cisplatin with etoposide/cisplatin in patients with previously untreated extensive-stage disease small-cell lung cancer. J Clin Oncol. 2006 May 1;24(13):2038-43. doi: 10.1200/JCO.2005.04.8595. PMID 16648503
- [Result] Hanna NH, Einhorn L, Sandler A, et al.: Randomized, phase III trial comparing irinotecan/cisplatin (IP) with etoposide/cisplatin (EP) in patients (pts) with previously untreated, extensive-stage (ES) small cell lung cancer (SCLC). [Abstract] Proceedings of the American Society of Clinical Oncology 23 (Suppl 16): A-LBA7004, 622s, 2005.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cisplatin + Irinotecan | Cisplatin + Etoposide
Started | 336 | 335
Completed | 194 | 217
Not Completed | 142 | 118
Not completed — Ineligible | 12 | 8
Not completed — Not treated | 7 | 2
Not completed — Adverse Event | 55 | 50
Not completed — Lack of Efficacy | 32 | 29
Not completed — Death | 10 | 10
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Other | 21 | 16

BASELINE CHARACTERISTICS:
Population: Eleven ineligible patients on the cisplatin + irinotecan arm, and eight ineligible patients on the cisplatin + etoposide arm were excluded from the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cisplatin + Irinotecan | Cisplatin + Etoposide | Total
Number analyzed (Participants) | 324 | 327 | 651
Age, Continuous [Median (Full Range); unit: years] | 62 [22 to 85] | 63 [35 to 88] | 62 [22 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136 | 145 | 281
  Male | 188 | 182 | 370
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 7 | 14
  Not Hispanic or Latino | 289 | 288 | 577
  Unknown or Not Reported | 28 | 32 | 60
Race/Ethnicity, Customized [Number; unit: particpants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 18 | 32
  White | 300 | 304 | 604
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 2 | 4 | 6

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival was defined as the duration between the date of randomization( enrollment) and the date of death due to any cause. Patients last known to be alive were censored at the date of last contact.
Time Frame: Weekly while on treatment, then every 3 months for first year, then every 6 months unitl a maximum of 3 years from enrollment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cisplatin + Irinotecan | Cisplatin + Etoposide
Number analyzed (Participants) | 324 | 327
Months | 9.9 [9.2 to 11.1] | 9.1 [8.4 to 9.9]

2. Secondary Outcome: Progression-free Survival
Description: Progression-Free Survival was defined as the duration from the date of randomization (enrollment) until the date of documentation of progression as defined by RECIST (a 20% increase over nadir in the sum of longest diameters of target lesions, clear progression of a non-target lesion in the opinion of the treating investigator, appearance of new lesions, or symptomatic deterioration) or death due to any cause. Patients last known to be alive and without evidence of progression were censored at the date of last contact.
Time Frame: Every 6 weeks until disease progression or a maximum of 3 years from the date of enrollment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cisplatin + Irinotecan | Cisplatin + Etoposide
Number analyzed (Participants) | 324 | 327
months | 5.7 [5.1 to 6.1] | 5.2 [4.9 to 5.5]

3. Secondary Outcome: Confirmed and Unconfirmed Complete and Partial Responses.
Description: Patients underwent chest CT/MRI every 6 weeks while on treatment and tumor response was evaluated by RECIST in the subset of patients with at least one target lesion at baseline. A target lesion was defined as a lesion with a longest diameter of at least 2 cm ( or at least 1 cm if by spiral CT). A complete response (CR) was defined as the disappearance of all disease, including non-target lesions. A partial response (PR) was defined as a 30% or greater decrease in the sum of the longest diameters. Confirmation of a CR or PR was defined as a second determination of CR or PR at least 4 weeks after the first determination.
Time Frame: Every 6 weeks while on protocol treatment for a maximum of 12 weeks
Measure: Number; unit: participants
Arm/Group | Cisplatin + Irinotecan | Cisplatin + Etoposide
Number analyzed (Participants) | 324 | 327
participants | 197 | 190

4. Secondary Outcome: Number of Patients With a Given Type and Grade of Adverse Event.
Description: Only adverse events that are possibly, probably or definitely related to study drug are reported. Only patients who received protocol treatment and were assessed for adverse events are included.
Time Frame: Every 4 weeks while subject on protocol treatment for a maximum of 12 weeks.
Population: Eligible patients who received protocol treatment.
Measure: Number; unit: Participants
Arm/Group | Cisplatin + Irinotecan | Cisplatin + Etoposide
Number analyzed (Participants) | 321 | 327
Participants
  ARDS | 0 | 1
  Abdominal pain/cramping | 8 | 8
  Acidosis | 2 | 1
  Alkaline phosphatase increase | 2 | 2
  Allergic reaction | 0 | 2
  Anal incontinence | 0 | 1
  Anemia | 19 | 40
  Anorexia | 36 | 17
  Anxiety/agitation | 0 | 1
  Apnea | 1 | 0
  Arrhythmia, NOS | 0 | 1
  Arthralgia | 0 | 1
  Ataxia (incoordination) | 1 | 2
  Bilirubin increase | 1 | 1
  Blurred vision | 0 | 1
  Bone pain | 8 | 6
  Cardiac ischemia/infarction | 1 | 2
  Cardiovascular-other | 1 | 1
  Cataract | 1 | 0
  Cerebrovascular ischemia | 1 | 7
  Chest pain,not cardio or pleur | 4 | 2
  Colitis | 2 | 1
  Confusion | 3 | 4
  Constipation/bowel obstruction | 4 | 4
  Creatinine increase | 9 | 7
  Dehydration | 54 | 27
  Delusions | 1 | 0
  Depression | 1 | 1
  Diarrhea without colostomy | 61 | 9
  Dizziness/light headedness | 2 | 4
  Dyspepsia/heartburn | 1 | 0
  Dyspnea | 27 | 21
  Edema | 1 | 1
  Epistaxis | 0 | 1
  Erythema multiforme/blistering | 0 | 1
  Esophagitis/dysphagia | 2 | 3
  Fatigue/malaise/lethargy | 45 | 35
  Febrile neutropenia | 11 | 33
  Fever without neutropenia | 1 | 0
  Flu-like symptoms-other | 2 | 2
  GGT increase | 0 | 1
  GI Mucositis, NOS | 0 | 2
  GI-other | 1 | 1
  GU-other | 2 | 0
  Gastric ulcer | 0 | 1
  Gastritis | 0 | 1
  Headache | 2 | 1
  Hematemesis | 0 | 1
  Hematologic-other | 1 | 0
  Hemorrhage-other | 0 | 1
  Hyperglycemia | 12 | 17
  Hyperkalemia | 3 | 1
  Hypermagnesemia | 1 | 0
  Hypernatremia | 1 | 2
  Hypertension | 2 | 4
  Hyperuricemia | 1 | 2
  Hypoalbuminemia | 2 | 7
  Hypocalcemia | 6 | 8
  Hypoglycemia | 2 | 3
  Hypokalemia | 19 | 21
  Hypomagnesemia | 3 | 7
  Hyponatremia | 38 | 28
  Hypophosphatemia | 7 | 5
  Hypotension | 14 | 8
  Hypoxia | 7 | 6
  Ileus | 2 | 0
  Infection w/o 3-4 neutropenia | 12 | 13
  Infection with 3-4 neutropenia | 20 | 24
  Infection, unk ANC | 2 | 3
  Inner ear-hearing loss | 1 | 4
  Insomnia | 1 | 2
  Joint,muscle,bone-other | 0 | 1
  LVEF decrease/CHF | 1 | 0
  Leukopenia | 57 | 109
  Lipase increase | 1 | 0
  Lung-other | 0 | 2
  Lymphopenia | 8 | 9
  Melena/ GI bleeding | 1 | 0
  Metabolic-other | 1 | 0
  Mood/consciousness change, NOS | 0 | 1
  Muscle weakness (not neuro) | 4 | 3
  Myalgia | 1 | 3
  Nausea | 46 | 35
  Neuro-other | 0 | 1
  Neutropenia/granulocytopenia | 108 | 224
  PRBC transfusion | 36 | 62
  Pain-other | 3 | 7
  Personality/behavioral change | 1 | 0
  Platelet transfusion | 1 | 13
  Pneumonitis/infiltrates | 4 | 2
  Pneumothorax | 0 | 1
  Prothrombin time increase | 3 | 2
  Pruritus | 0 | 1
  RT-pain | 0 | 1
  Rash/desquamation | 0 | 3
  Renal failure | 4 | 7
  Reportable adverse event, NOS | 1 | 1
  Respiratory infect w/ neutrop | 3 | 1
  Respiratory infect w/o neutrop | 3 | 1
  Respiratory infection, unk ANC | 1 | 0
  SGOT (AST) increase | 3 | 4
  SGPT (ALT) increase | 3 | 3
  SIADH | 2 | 3
  Second primary | 2 | 0
  Seizures | 2 | 1
  Sensory neuropathy | 1 | 1
  Sinus tachycardia | 0 | 1
  Somnolence/consciousness loss | 2 | 1
  Stomatitis/pharyngitis | 1 | 0
  Supraventricular arrhythmia | 3 | 0
  Syncope | 5 | 7
  Thrombocytopenia | 13 | 52
  Thrombosis/embolism | 8 | 15
  Thrombotic microangiopathy | 1 | 0
  Tumor lysis syndrome | 2 | 2
  Ureteral obstruction | 0 | 1
  Urinary electrolyte wasting | 0 | 1
  Urinary retention | 1 | 1
  Urinary tr infect w/ neutrop | 1 | 0
  Ventricular arrhythmia | 1 | 1
  Voice change/stridor/larynx | 2 | 0
  Vomiting | 34 | 30
  Weakness (motor neuropathy) | 1 | 0
  Weight loss | 3 | 1

ADVERSE EVENTS:
Time Frame: Patients were evaluated for adverse events prior to the beginning of each cycle of treatment, approximately every 4 weeks, for up to a maximum of 4 cycles (16 weeks).
Description: Eligible patients who received at least one dose of treatment were included in the analysis of adverse events.
Arm/Group | Cisplatin + Irinotecan | Cisplatin + Etoposide
Serious Adverse Events (participants affected / at risk) | 107/321 | 31/327
Other Adverse Events (participants affected / at risk) | 314/321 | 317/327
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cisplatin + Irinotecan (N=321) | Cisplatin + Etoposide (N=327)
Anemia (Blood and lymphatic system disorders) | 3 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 0
PRBC transfusion (Blood and lymphatic system disorders) | 1 | 0
Platelet transfusion (Blood and lymphatic system disorders) | 2 | 0
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 | 0
Cardiac ischemia/infarction (Cardiac disorders) | 0 | 1
Cardiovascular-other (Cardiac disorders) | 2 | 0
LVEF decrease/CHF (Cardiac disorders) | 1 | 0
Supraventricular arrhythmia (Cardiac disorders) | 4 | 0
Ventricular arrhythmia (Cardiac disorders) | 3 | 1
Abdominal pain/cramping (Gastrointestinal disorders) | 2 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation/bowel obstruction (Gastrointestinal disorders) | 1 | 0
Diarrhea without colostomy (Gastrointestinal disorders) | 29 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 8 | 0
Rectal bleeding/hematochezia (Gastrointestinal disorders) | 0 | 1
Stomatitis/pharyngitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 13 | 0
Edema (General disorders) | 2 | 0
Fatigue/malaise/lethargy (General disorders) | 11 | 0
Flu-like symptoms-other (General disorders) | 11 | 6
Pain-other (General disorders) | 2 | 0
Reportable adverse event, NOS (General disorders) | 1 | 4
Infection w/o 3-4 neutropenia (Infections and infestations) | 6 | 1
Infection with 3-4 neutropenia (Infections and infestations) | 8 | 6
Infection, unk ANC (Infections and infestations) | 1 | 0
Respiratory infect w/ neutrop (Infections and infestations) | 2 | 1
Respiratory infect w/o neutrop (Infections and infestations) | 2 | 0
Respiratory infection, unk ANC (Infections and infestations) | 2 | 0
Urinary tr infect w/ neutrop (Infections and infestations) | 1 | 0
Abnormal troponin I (cTnI) (Investigations) | 1 | 1
Amylase increase (Investigations) | 1 | 0
CPK increase (Investigations) | 1 | 0
Creatinine increase (Investigations) | 9 | 1
Leukopenia (Investigations) | 5 | 0
Lipase increase (Investigations) | 1 | 0
Neutropenia/granulocytopenia (Investigations) | 19 | 0
Prothrombin time increase (Investigations) | 2 | 0
SIADH (Investigations) | 1 | 0
Thrombocytopenia (Investigations) | 1 | 1
Weight loss (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 7 | 0
Dehydration (Metabolism and nutrition disorders) | 33 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalemia (Metabolism and nutrition disorders) | 5 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 11 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Chest pain,not cardio or pleur (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint,muscle,bone-other (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscle weakness (not neuro) (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia/arthralgia, NOS (Musculoskeletal and connective tissue disorders) | 1 | 0
Second primary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ataxia (incoordination) (Nervous system disorders) | 1 | 0
CNS hemorrhage (Nervous system disorders) | 1 | 0
Cerebrovascular ischemia (Nervous system disorders) | 3 | 1
Dizziness/vertigo, NOS (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Neuropathic pain (Nervous system disorders) | 1 | 0
Seizures (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 0
Weakness (motor neuropathy) (Nervous system disorders) | 0 | 1
Anxiety/agitation (Psychiatric disorders) | 1 | 0
Confusion (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Hallucinations (Psychiatric disorders) | 1 | 0
Mood/consciousness change, NOS (Psychiatric disorders) | 2 | 0
Personality/behavioral change (Psychiatric disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 1
Urinary electrolyte wasting (Renal and urinary disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
ARDS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 | 3
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Pneumonitis/infiltrates (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypotension (Vascular disorders) | 9 | 0
Peripheral arterial ischemia (Vascular disorders) | 1 | 0
Thrombosis/embolism (Vascular disorders) | 10 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cisplatin + Irinotecan (N=321) | Cisplatin + Etoposide (N=327)
Anemia (Blood and lymphatic system disorders) | 214 | 240
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 34
PRBC transfusion (Blood and lymphatic system disorders) | 35 | 62
Ear-other (Ear and labyrinth disorders) | 0 | 18
Inner ear-hearing loss (Ear and labyrinth disorders) | 0 | 30
Abdominal pain/cramping (Gastrointestinal disorders) | 64 | 45
Constipation/bowel obstruction (Gastrointestinal disorders) | 73 | 99
Diarrhea without colostomy (Gastrointestinal disorders) | 182 | 85
Dyspepsia/heartburn (Gastrointestinal disorders) | 18 | 26
Nausea (Gastrointestinal disorders) | 215 | 228
Stomatitis/pharyngitis (Gastrointestinal disorders) | 31 | 38
Vomiting (Gastrointestinal disorders) | 132 | 142
Edema (General disorders) | 51 | 53
Fatigue/malaise/lethargy (General disorders) | 233 | 246
Pain-other (General disorders) | 32 | 46
Infection w/o 3-4 neutropenia (Infections and infestations) | 43 | 43
Infection with 3-4 neutropenia (Infections and infestations) | 0 | 18
Alkaline phosphatase increase (Investigations) | 50 | 59
Creatinine increase (Investigations) | 45 | 66
Leukopenia (Investigations) | 162 | 208
Lymphopenia (Investigations) | 0 | 23
Neutropenia/granulocytopenia (Investigations) | 175 | 255
SGOT (AST) increase (Investigations) | 41 | 35
SGPT (ALT) increase (Investigations) | 40 | 37
Thrombocytopenia (Investigations) | 79 | 167
Weight loss (Investigations) | 98 | 85
Anorexia (Metabolism and nutrition disorders) | 133 | 133
Dehydration (Metabolism and nutrition disorders) | 76 | 71
Hyperglycemia (Metabolism and nutrition disorders) | 87 | 78
Hyperkalemia (Metabolism and nutrition disorders) | 17 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 51 | 60
Hypocalcemia (Metabolism and nutrition disorders) | 55 | 60
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 17
Hypokalemia (Metabolism and nutrition disorders) | 49 | 50
Hypomagnesemia (Metabolism and nutrition disorders) | 43 | 47
Hyponatremia (Metabolism and nutrition disorders) | 68 | 72
Bone pain (Musculoskeletal and connective tissue disorders) | 23 | 33
Chest pain,not cardio or pleur (Musculoskeletal and connective tissue disorders) | 17 | 0
Muscle weakness (not neuro) (Musculoskeletal and connective tissue disorders) | 18 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 24 | 20
Dizziness/light headedness (Nervous system disorders) | 26 | 29
Headache (Nervous system disorders) | 25 | 28
Sensory neuropathy (Nervous system disorders) | 45 | 52
Taste disturbance (Nervous system disorders) | 23 | 25
Anxiety/agitation (Psychiatric disorders) | 17 | 0
Depression (Psychiatric disorders) | 17 | 0
Insomnia (Psychiatric disorders) | 28 | 29
Cough (Respiratory, thoracic and mediastinal disorders) | 48 | 43
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 106 | 98
Alopecia (Skin and subcutaneous tissue disorders) | 132 | 204
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 | 30
Hypotension (Vascular disorders) | 21 | 29
Thrombosis/embolism (Vascular disorders) | 0 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No